CLINICAL TRIAL: NCT00798915
Title: Restoration of the GIP-mediated Incretin Effect in Persons With Type 2 Diabetes Mellitus
Brief Title: Study of the Effects of Xenin-25 in Humans With and Without Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 08-0861A; 1RC1DK086163-01 (NIH)
Record Dates: First submitted 2008-11-24; First posted 2008-11-26 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Diabetes
Keywords: Diabetes; Blood Sugar; Xenin-25; GIP; Insulin
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Incretins; xenin 25

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal Glucose Tolerance (Experimental): Healthy individuals exhibiting plasma glucose levels less than 140mg/dl two hours after ingestion of 75-g of glucose.
  Interventions: Drug: Placebo; Drug: Glucose-dependent Insulinotropic Polypeptide (GIP); Drug: Xenin-25; Drug: Glucose-dependent Insulinotropic Polypeptide plus Xenin-25
- Impaired Glucose Tolerance (Experimental): Healthy individuals exhibiting plasma glucose levels between 140 and 199 mg/dl two hours after ingestion of 75-g of glucose.
  Interventions: Drug: Placebo; Drug: Glucose-dependent Insulinotropic Polypeptide (GIP); Drug: Xenin-25; Drug: Glucose-dependent Insulinotropic Polypeptide plus Xenin-25
- Type 2 diabetes mellitus (Experimental): Healthy individuals exhibiting plasma glucose levels greater than 150 mg/dL under fasting conditions OR greater than 199 mg/dl two hours after ingestion of 75-g of glucose.
  Interventions: Drug: Placebo; Drug: Glucose-dependent Insulinotropic Polypeptide (GIP); Drug: Xenin-25; Drug: Glucose-dependent Insulinotropic Polypeptide plus Xenin-25

INTERVENTIONS:
Drug: Placebo — Intravenous infusion of 1% human albumin in normal saline
  Other Names: Vehicle alone
Drug: Glucose-dependent Insulinotropic Polypeptide (GIP) — Intravenous infusion of GIP (4 pmoles x kg-1 x min-1) in 1% human albumin in normal saline
  Other Names: GIP
Drug: Xenin-25 — Intravenous infusion of xenin-25 (4 pmoles x kg-1 x min-1) in 1% human albumin in normal saline
  Other Names: Xenin
Drug: Glucose-dependent Insulinotropic Polypeptide plus Xenin-25 — Intravenous infusion of GIP plus xenin-25 (4 pmoles each x kg-1 x min-1) in 1% human albumin in normal saline
  Other Names: GIP plus Xenin

SUMMARY:
An intestinal hormone called Glucose-dependent Insulinotropic Polypeptide (GIP) is released into the blood immediately after ingestion of a meal and plays an important role in regulating blood sugar levels. However, GIP is not active in persons with type 2 diabetes mellitus (T2DM) which is also known as adult onset or non-insulin-dependent diabetes. This study is being conducted to determine whether a hormone called xenin-25 can restore the activity of GIP in persons with T2DM.

DETAILED DESCRIPTION:
Each eligible participant will be administered an oral glucose tolerance test so he/she can be assigned to the group with "normal glucose tolerance", "impaired glucose tolerance" (between normal and diabetic), or type 2 diabetes mellitus. Each study subject will then be administered a graded glucose infusion (GGI) on 4 separate occasions. For the GGI, an intravenous glucose infusion will be started at a rate of 1 mg x kg-1 x min-1 for 40 min, followed by 2, 3, 4, 6, and 8 mg x kg-1 x min-1 (40 min for each step). A primed-continuous infusion of vehicle alone, GIP alone, xenin-25 alone, or the combination of GIP plus xenin-25 (each peptide at a dose of 4 pmoles x kg-1 x min-1) will be initiated at the same time the glucose infusion is started. Blood samples will be collected before and during the GGI for the measurement of glucose, insulin, C-peptide, glucagon, GIP and xenin-25 levels.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be able to consent for their own participation (no mental impairment affecting cognition or willingness to follow study instructions).
* Healthy volunteers with no clinical evidence of T2DM.
* Otherwise healthy volunteers that have impaired glucose tolerance.
* Otherwise healthy volunteers with diet controlled T2DM.
* Otherwise healthy volunteers with T2DM that take oral agents only if the subject's pre-existing oral anti-diabetic agents can be safely discontinued for 48-hours.
* Persons with HbA1c less than 9%.
* Women of childbearing potential must be currently taking/using an acceptable method of birth control. A pregnancy test will be done at the beginning of each visit. Any woman with a positive pregnancy test will be removed from the study.
* Willingness to complete all required visits.

Exclusion Criteria:

* Lacks cognitive ability to sign the consent or follow the study directions.
* Women unwilling to use an acceptable method of contraception during the course of the study, or who are currently breast-feeding.
* Any subject whose screening HbA1c is >9.0%.
* Type 2 diabetes requiring the use of supplemental insulin at home.
* Volunteers with a history of Acute Pancreatitis.
* Volunteers with a history of cancer (except for skin cancer).
* Volunteer with a history of Chronic Pancreatitis and/or risk factors for chronic pancreatitis including hypertriglyceridemia (triglycerides >400mg/ml) hypercalcemia (blood calcium level >11.md/dl) and/or the presence of gallstones.
* Volunteers with a history of gastrointestinal disorders, particularly related to gastric motility/emptying such as gastric bypass, documented gastro-paresis in diabetic volunteers.
* Subjects taking medications known to affect glucose tolerance.
* Hematocrit from the lab is below 33% (or if the finger stick hemoglobin measured with the HemoCue 201+ is <11.2% mg/dlL).
* Diabetics that have the potential to have a low blood sugar without them being aware that their blood sugar is low (hypoglycemia unawareness).
* Significant systemic illness including heart, kidney, inflammatory, liver, or malignant disease requiring medications.
* Subjects will be excluded if their liver or kidney function is outside the upper limits of normal by > 3%. Total Bilirubin levels should be <2.
* Subjects unwilling to allow the use of human albumin in the preparation of the peptides.
* Unwillingness to allow blood glucose level adjustment (if needed) with IV insulin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The effects of GIP, xenin-25, or a combination of GIP plus xenin-25 on insulin secretion and blood glucose levels | 5 years

SECONDARY OUTCOMES:
The effects of xenin-25 on GIP action in persons with type 2 diabetes | 5yrs

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Reeds, MD, Principal Investigator — Washington University School of Medicine; Burton Wice, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Chowdhury S, Wang S, Patterson BW, Reeds DN, Wice BM. The combination of GIP plus xenin-25 indirectly increases pancreatic polypeptide release in humans with and without type 2 diabetes mellitus. Regul Pept. 2013 Nov 10;187:42-50. doi: 10.1016/j.regpep.2013.10.003. Epub 2013 Oct 29. PMID 24183983
- [Result] Wice BM, Reeds DN, Tran HD, Crimmins DL, Patterson BW, Dunai J, Wallendorf MJ, Ladenson JH, Villareal DT, Polonsky KS. Xenin-25 amplifies GIP-mediated insulin secretion in humans with normal and impaired glucose tolerance but not type 2 diabetes. Diabetes. 2012 Jul;61(7):1793-800. doi: 10.2337/db11-1451. Epub 2012 Apr 20. PMID 22522617